CLINICAL TRIAL: NCT04305990
Title: Feasibility and Comfort of a Nasal Demand-Driven Method for Gas Delivery in a Dental Setting
Brief Title: Demand-Driven Method for Gas Delivery in a Dental Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: O-Two Medical Technologies (Unknown)
Responsible Party: Principal Investigator, Carilynne Yarascavitch, Assistant Professor, Specialty Program Director, Dental Anaesthesia, Faculty of Dentistry, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 00038876
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Nitrous Oxide; Dentistry; Drug Delivery System; Comfort; Feasibility; Drug Administration, Inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: The study design is a within-subjects, single-blinded, randomized controlled trial. Each participant will receive both the free-flow (FF) and demand-driven (DD) gas delivery methods in a randomized sequence.
Who Masked: Participant
Masking Description: Participants will not be told the order the gas flow delivery method (DD or FF) they will be receive. To assist with masking participants, the same device and nasal hood will be used throughout, they will be told to face forward away from the device and device display, which indicates the setting of the gas flow. It will not be feasible to blind the researcher as the researcher will need to change the device setting (FF or DD).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Demand-driven delivery followed by free-flow delivery (Experimental): Participants will inspire 100% oxygen through their nose with the gas delivery device set to a demand-driven delivery setting through a nasal hood for 2 minutes followed by inspiration of 100% oxygen through their nose with the gas delivery device set to a free-flow delivery setting through a nasal hood for 2 minutes.
  Interventions: Device: Demand-driven delivery method; Device: Free-flow delivery method
- Free-flow delivery followed by demand-driven delivery (Experimental): Participants will inspire 100% oxygen through their nose with the gas delivery device set to a free-flow delivery setting through a nasal hood for 2 minutes followed by inspiration of 100% oxygen through their nose with the gas delivery device set to a free-flow delivery setting through a nasal hood for 2 minutes.
  Interventions: Device: Demand-driven delivery method; Device: Free-flow delivery method

INTERVENTIONS:
Device: Demand-driven delivery method — The gas delivery device is set to the demand-driven setting. Patients must inspire through their nose to trigger the flow of gas.
Device: Free-flow delivery method — The gas delivery device is set to a free-flow setting. Gas flows through the system at a rate determined by the operator. Standard flow rate is 6 liters per minute. Patients do not need to inspire through their nose to trigger the flow of gas.

SUMMARY:
This study compares two methods of gas delivery in a dental setting: 1) demand-driven (DD) and 2) free-flow (FF).

Nitrous oxide and oxygen sedation (NOS) is a common form of minimal sedation for adult and paediatric patients undergoing dental procedures. In order for NOS devices to be utilized during dental treatment, dentists must be able to provide gas flow to the patient, and subsequently scavenge used and unused gasses. Gas delivery is via a nasal mask, since the oral cavity must be accessible to the dentist throughout treatment.

Current devices for NOS in the dental setting utilize a free-flow gas method, where nitrous oxide and oxygen are released continuously from their tanks. The flow rate is set by the dentist according to the patient's minute ventilation needs, and unused and exhaled gasses are scavenged via the nasal mask. The demand-driven gas flow method, where inspiration triggers gas flow, has been used successfully in other medical settings, such as in obstetrics, medical emergencies, and for patients with chronic obstructive pulmonary disease. However, in these settings the mask used covers both the nose and mouth, and patients can trigger the demand-driven method through inspiration of the nose or mouth. The demand-driven gas flow method has a significant gas-sparing advantage over the free-flow method. With a demand-driven method, the patient dictates the flow rate and gas is only delivered when they are inspiring, compared to the free-flow method which provide gas flow throughout inspiration and expiration. However, the demand-driven method have not been studied in a dental setting where flow can only be triggered through the nose. It is therefore unknown whether it is feasible or comfortable for patients to trigger a demand-driven method nasally when their mouth is open during dental treatment.

This study will aim to assess the feasibility and comfort of a nasal demand-driven gas delivery method utilizing 100% oxygen in healthy, adult participants in a simulated dental setting. If the device is feasible and comfortable with 100% oxygen in a simulated dental setting, future research can be conducted to assess its use for NOS for dental treatment.

DETAILED DESCRIPTION:
The study design is a within-subjects, single-blinded, randomized control trial. Participants will be randomzied to inspire 100% oxygen through their nose utilizing a demand-driven (DD) gas delivery method and a free-flow (FF) gas delivery method for 2 minutes each in a simulated dental setting.

The study will take place at the University of Toronto's Faculty of Dentistry Children's Clinic. Participants will be positioned supine in the dental chair. A child size, rubber bite block will be inserted with an attached capnography device to measure end-tidal carbon dioxide at the mouth. A double-mask nasal hood with disposable insert will be placed on the participant's nose. The participant will be instructed to breathe through their mouth for 1 minute. Baseline respiratory rate and presence/absence of end tidal carbon dioxide at the mouth will be obtained through the capnograph and recorded. The presence of carbon dioxide at baseline during mouth breathing will confirm that the capnograph is able to measure end-tidal carbon dioxide at the mouth.

The researcher will then open the envelope with the randomization plan for the participant and will indicate whether they will receive the FF or DD gas delivery method first. The gas delivery device will be attached to the nasal hood, and set to either DD or FF gas delivery method. Once the device is connected, the participant will be instructed to breathe through their nose for 2 minutes. During this time, respiratory rate, presence/absence of end tidal carbon dioxide at the mouth, and oxygen flow rate per minute will be observed and recorded. The absence of end-tidal carbon dioxide at the mouth during this testing phase will provide a verifiable measure that patients are breathing through their nose. After 2 minutes, the flow will be stopped and the bite block removed. The participant will be instructed to breathe through their mouth. The participant will then complete the VAS on comfort of breathing through their nose during the first gas flow delivery method. The bite block will then be reinserted, and the flow resumed using the second gas flow delivery method for 2 minutes. During this time, respiratory rate, presence/absence of end tidal carbon dioxide at the mouth, and oxygen flow rate per minute will be observed and recorded. After 2 minutes, the gas flow will once again be stopped and the bite block removed. The participant will be instructed to complete the VAS on comfort of breathing through their nose. The nasal hood will be removed. The participant will be debriefed to the order of gas flow received (DD or FF first) and the participant will then be dismissed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be adults, 18 years of age or older.
2. Participants must be ASA I (a normal, healthy patient) or ASA II (a patient with mild systemic disease).

Exclusion Criteria:

1. Participants who are ASA III (a patient with a severe systemic disease that is not life-threatening) or higher.
2. Participants who indicate they are claustrophobic.
3. Participants with nasal obstruction of both nostrils.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Comfort of the demand-driven gas delivery mechanism | Assessed immediately after breathing through each mechanism for 2 minutes
  To assess patient comfort of breathing through their nose with the demand-driven gas delivery method vs the free-flow method. In order to assess comfort, the patient will report perceived comfort on a 100mm visual analog scale immediately after each device is turned on. We will test for non-inferiority in comfort of the demand-driven as compared to the free-flow delivery method.
Feasibility of the demand-driven gas delivery mechanism | Procedure (Assessed for the duration of time when the patient is breathing from either delivery system)
  To assess whether it is feasible for participants to inspire 100% oxygen through a nasal hood when utilizing a demand-driven gas delivery mechanism when their mouth is open, in a simulated dental setting. In order to assess feasibility, we will monitor for the presence or absence end-tidal carbon dioxide at the mouth to confirm whether the patient is breathing through their nose or mouth. Absence of carbon dioxide at the mouth indicates the patient was able to trigger the mechanism and breathe through their nose.

CONTACTS AND LOCATIONS:
Overall Officials: Carilynne Yarascavitch, BSc DDS MSc, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Faculty of Dentistry, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson S, Gosnell ES. Survey of American Academy of Pediatric Dentistry on Nitrous Oxide and Sedation: 20 Years Later. Pediatr Dent. 2016 Oct 15;38(5):385-392. PMID 28206894
- [Background] Malamed SF, Clark MS. Nitrous oxide-oxygen: a new look at a very old technique. J Calif Dent Assoc. 2003 May;31(5):397-403. PMID 12839232
- [Background] Becker DE, Rosenberg M. Nitrous oxide and the inhalation anesthetics. Anesth Prog. 2008 Winter;55(4):124-30; quiz 131-2. doi: 10.2344/0003-3006-55.4.124. PMID 19108597
- [Background] Clark MS, Brunick A. Handbook of Nitrous Oxide and Oxygen Sedation. 5th Edition ed: Elsevier Health Sciences; 2019.
- [Background] Tiep BL, Nicotra MB, Carter R, Phillips R, Otsap B. Low-concentration oxygen therapy via a demand oxygen delivery system. Chest. 1985 May;87(5):636-8. doi: 10.1378/chest.87.5.636. PMID 3921316
- [Background] van der Kooy J, De Graaf JP, Kolder ZM, Witters KD, Fitzpatrick E, Duvekot JJ, Dons-Sinke IJ, Steegers EA, Bonsel GJ. A newly developed scavenging system for administration of nitrous oxide during labour: safe occupational use. Acta Anaesthesiol Scand. 2012 Aug;56(7):920-5. doi: 10.1111/j.1399-6576.2012.02668.x. Epub 2012 Mar 7. PMID 22404276
- [Background] Dallal GD. Randomization.com [updated July 15, 2008. Available from: ⟨http://www.randomization.com/⟩.
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Humphris GM, Morrison T, Lindsay SJ. The Modified Dental Anxiety Scale: validation and United Kingdom norms. Community Dent Health. 1995 Sep;12(3):143-50. PMID 7584581
- [Background] Humphris GM, Dyer TA, Robinson PG. The modified dental anxiety scale: UK general public population norms in 2008 with further psychometrics and effects of age. BMC Oral Health. 2009 Aug 26;9:20. doi: 10.1186/1472-6831-9-20. PMID 19709436
- [Background] Humphris G, Crawford JR, Hill K, Gilbert A, Freeman R. UK population norms for the modified dental anxiety scale with percentile calculator: adult dental health survey 2009 results. BMC Oral Health. 2013 Jun 24;13:29. doi: 10.1186/1472-6831-13-29. PMID 23799962
- [Background] King K, Humphris G. Evidence to confirm the cut-off for screening dental phobia using the Modified Dental Anxiety Scale. Soc sci dent. 2010;1(1):21-8.
- [Background] Hendrix JM, Garmon EH. American Society of Anesthesiologists Physical Status Classification System. 2025 Feb 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441940/ PMID 28722969